CLINICAL TRIAL: NCT04270838
Title: A Phase Ib/II Age De-escalation, Dose Escalation, Partially Randomised, Open-label Head-to-head Study of the Safety and Immunogenicity of the Candidate Rabies Vaccine ChAdOx2 RabG
Brief Title: A Phase Ib/II Study of the Safety and Immunogenicity of the Candidate Rabies Vaccine ChAdOx2 RabG
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Ifakara Health Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RAB002
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Rabies
Keywords: Vaccine
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Group AC1 (Adult low dose) (Experimental): Volunteers aged 18-45 years. Volunteers will receive a standalone dose of 2.5×10^10 vp ChAdOx2 RabG on D0. Volunteers will receive two doses of Rabies IRV as simulated post-exposure prophylaxis (SPEP), 14 days apart during the follow-up period. All participants will receive Verorab as a 4 site ID on SPEP+0, and Verorab as a 2 site ID on SPEP+14. Participants who return a virus neutralising antibody (VNA) result below 0.5IU/mL will be randomised (1:1 ratio) for the SPEP+0 visit to happen at the next available visit or at the final annual visit. Any participants who do not return a VNA result below 0.5IU/mL will have their SPEP+0 visit take place at the final annual visit.
  Interventions: Biological: ChAdOx2 RabG; Biological: Inactivated Rabies Vaccine
- Group AC2 (Adult high dose) (Experimental): Volunteers aged 18-45 years. Volunteers will receive a standalone dose of 5×10^10 vp ChAdOx2 RabG. Volunteers will receive two doses of Rabies IRV as simulated post-exposure prophylaxis (SPEP), 14 days apart during the follow-up period. All participants will receive Verorab as a 4 site ID on SPEP+0, and Verorab as a 2 site ID on SPEP+14. Participants who return a virus neutralising antibody (VNA) result below 0.5IU/mL will be randomised (1:1 ratio) for the SPEP+0 visit to happen at the next available visit or at the final annual visit. Any participants who do not return a VNA result below 0.5IU/mL will have their SPEP+0 visit take place at the final annual visit.
  Interventions: Biological: ChAdOx2 RabG; Biological: Inactivated Rabies Vaccine
- Group AC3 (Adult preferred dose) (Experimental): Volunteers aged 18-45 years. Volunteers will receive a preferred dose of ChAdOx2 RabG on D0. The adult preferred dose will be 2.5×10^10 vp OR 5×10^10 vp. Volunteers will receive two doses of Rabies IRV as simulated post-exposure prophylaxis (SPEP), 14 days apart during the follow-up period. All participants will receive Verorab as a 4 site ID on SPEP+0, and Verorab as a 2 site ID on SPEP+14. Participants who return a virus neutralising antibody (VNA) result below 0.5IU/mL will be randomised (1:1 ratio) for the SPEP+0 visit to happen at the next available visit or at the final annual visit. Any participants who do not return a VNA result below 0.5IU/mL will have their SPEP+0 visit take place at the final annual visit.
  Interventions: Biological: ChAdOx2 RabG; Biological: Inactivated Rabies Vaccine
- Group AV1 (Adult single-visit Verobab) (Experimental): Volunteers aged 18-45 years. Volunteers will receive Rabies IRV on D0. Volunteers will receive two further doses of Rabies IRV as simulated post-exposure prophylaxis (SPEP), 14 days apart during the follow-up period. All participants will receive Verorab as a 4 site ID on SPEP+0, and Verorab as a 2 site ID on SPEP+14. Participants who return a virus neutralising antibody (VNA) result below 0.5IU/mL will be randomised (1:1 ratio) for the SPEP+0 visit to happen at the next available visit or at the final annual visit. Any participants who do not return a VNA result below 0.5IU/mL will have their SPEP+0 visit take place at the final annual visit.
  Interventions: Biological: Inactivated Rabies Vaccine
- PC1a (Paediatric low dose) (Experimental): Volunteers aged 2-6 years. Volunteers will receive a standalone dose of 1×10^10 vp ChAdOx2 RabG on D0. Volunteers will receive two doses of Rabies IRV as simulated post-exposure prophylaxis (SPEP), 14 days apart during the follow-up period. All participants will receive Verorab as a 4 site ID on SPEP+0, and Verorab as a 2 site ID on SPEP+14. Participants who return a virus neutralising antibody (VNA) result below 0.5IU/mL will be randomised (1:1 ratio) for the SPEP+0 visit to happen at the next available visit or at the final annual visit. Any participants who do not return a VNA result below 0.5IU/mL will have their SPEP+0 visit take place at the final annual visit.
  Interventions: Biological: ChAdOx2 RabG; Biological: Inactivated Rabies Vaccine
- PC1b (Paediatric low dose) (Experimental): Volunteers aged 2-6 years. Volunteers will receive a half adult preferred dose of ChAdOx2 RabG on D0. The adult preferred dose will be 2.5×10^10 vp OR 5×10^10 vp. Volunteers will receive two doses of Rabies IRV as simulated post-exposure prophylaxis (SPEP), 14 days apart during the follow-up period. All participants will receive Verorab as a 4 site ID on SPEP+0, and Verorab as a 2 site ID on SPEP+14. Participants who return a virus neutralising antibody (VNA) result below 0.5IU/mL will be randomised (1:1 ratio) for the SPEP+0 visit to happen at the next available visit or at the final annual visit. Any participants who do not return a VNA result below 0.5IU/mL will have their SPEP+0 visit take place at the final annual visit.
  Interventions: Biological: ChAdOx2 RabG; Biological: Inactivated Rabies Vaccine
- PC2 (Paediatric high dose) (Experimental): Volunteers aged 2-6 years. Volunteers will receive a full adult preferred dose of ChAdOx2 RabG on D0. The adult preferred dose will be 2.5×10^10 vp OR 5×10^10 vp. Volunteers will receive two doses of Rabies IRV as simulated post-exposure prophylaxis (SPEP), 14 days apart during the follow-up period. All participants will receive Verorab as a 4 site ID on SPEP+0, and Verorab as a 2 site ID on SPEP+14. Participants who return a virus neutralising antibody (VNA) result below 0.5IU/mL will be randomised (1:1 ratio) for the SPEP+0 visit to happen at the next available visit or at the final annual visit. Any participants who do not return a VNA result below 0.5IU/mL will have their SPEP+0 visit take place at the final annual visit.
  Interventions: Biological: ChAdOx2 RabG; Biological: Inactivated Rabies Vaccine
- PC3 (Paediatric preferred dose) (Experimental): Volunteers aged 2-6 years. Volunteers will receive a paediatric preferred dose of ChAdOx2 RabG on D0. The paediatric preferred dose will be 50-100% of the adult preferred dose. Volunteers will receive two doses of Rabies IRV as simulated post-exposure prophylaxis (SPEP), 14 days apart during the follow-up period. All participants will receive Verorab as a 4 site ID on SPEP+0, and Verorab as a 2 site ID on SPEP+14. Participants who return a virus neutralising antibody (VNA) result below 0.5IU/mL will be randomised (1:1 ratio) for the SPEP+0 visit to happen at the next available visit or at the final annual visit. Any participants who do not return a VNA result below 0.5IU/mL will have their SPEP+0 visit take place at the final annual visit.
  Interventions: Biological: ChAdOx2 RabG; Biological: Inactivated Rabies Vaccine
- PV1 (Paediatric single-visit Verobab) (Experimental): Volunteers aged 2-6 years. Volunteers will receive Rabies IRV (Verorab) as a 2 site ID on D0. Volunteers will receive two further doses of Rabies IRV as simulated post-exposure prophylaxis (SPEP), 14 days apart during the follow-up period. All participants will receive Verorab as a 4 site ID on SPEP+0, and Verorab as a 2 site ID on SPEP+14. Participants who return a virus neutralising antibody (VNA) result below 0.5IU/mL will be randomised (1:1 ratio) for the SPEP+0 visit to happen at the next available visit or at the final annual visit. Any participants who do not return a VNA result below 0.5IU/mL will have their SPEP+0 visit take place at the final annual visit.
  Interventions: Biological: Inactivated Rabies Vaccine
- PV2 (Paediatric two-visit Verobab) (Experimental): Volunteers aged 2-6 years. Volunteers will receive Rabies IRV (Verorab) as a 2 site ID on D0. Volunteers will receive two further doses of Rabies IRV as simulated post-exposure prophylaxis (SPEP), 14 days apart during the follow-up period. All participants will receive Verorab as a 4 site ID on SPEP+0, and Verorab as a 2 site ID on SPEP+14. Participants who return a virus neutralising antibody (VNA) result below 0.5IU/mL will be randomised (1:1 ratio) for the SPEP+0 visit to happen at the next available visit or at the final annual visit. Any participants who do not return a VNA result below 0.5IU/mL will have their SPEP+0 visit take place at the final annual visit.
  Interventions: Biological: Inactivated Rabies Vaccine

INTERVENTIONS:
Biological: ChAdOx2 RabG — Single dose of ChAdOx2 RabG at different concentrations: 1x10^10 and 5x10^10
  Arms: Group AC1 (Adult low dose); Group AC2 (Adult high dose); Group AC3 (Adult preferred dose); PC1a (Paediatric low dose); PC1b (Paediatric low dose); PC2 (Paediatric high dose); PC3 (Paediatric preferred dose)
Biological: Inactivated Rabies Vaccine — A complete pre-exposure prophylactic course of an existing rabies vaccine, ≥2.5 international units
  Other Names: Verorab

SUMMARY:
This is a Phase Ib/II, open-label, head-to-head, age de-escalation dose-escalation, partially randomized trial to study the safety and immunogenicity of the candidate rabies vaccine ChAdOx2 RabG in healthy adults (age 18-45 years) and young children (age 2-6 years). ChAdOx2 RabG will be administered intramuscularly and licensed rabies vaccine will be given by intradermal injection.

DETAILED DESCRIPTION:
A total of 120 participants will be recruited into 10 groups in Bagamoyo, Tanzania. The duration of the entire study will be up to 5.5 years per participant from the time of first vaccination. ChAdOx2 RabG will be administered intramuscularly and licensed rabies vaccine (Verorab) will be given by intradermal injection at two to four anatomical sites (deltoids, thighs or suprascapular areas).

All participants, regardless of which vaccine they receive at the start of the study, will receive a course of a licenced rabies vaccine (Verorab) during or at the end of the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Adult groups: Healthy male or female adults aged 18-45 years at the time of enrolment with signed consent.
* Adult groups (Female only participants): Must be non-pregnant (as demonstrated by a negative urine pregnancy test) and willing to use an effective form of contraception. Or if they agree to an extended period of follow-up of up to 5.5 years, use an effective form of contraception during the first year of enrolment in the study).
* Paediatric groups: Healthy male or female young children aged 2-6 years at the time of enrolment with signed consent obtained from parents or guardians.
* Paediatric groups: completion of the Expanded Programme on Immunisation (EPI) at least 6 months prior to study enrolment.
* Planned long-term (at least 61 months from the date of the first vaccination) or permanent residence in Bagamoyo town.
* Adults with a Body Mass Index (BMI) 18 to 35 Kg/m2; or young children with Z-score of weight-for-age within ±2SD.
* Correctly answer all 10 questions on the protocol and study procedures understanding questionnaire within 2 attempts.

Exclusion Criteria:

* Clinically significant congenital abnormalities as judged by the PI or other delegated individual.
* Clinically significant history of skin disorder, allergy, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease and neurological illness which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data as judged by the PI or other delegated individual.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* Any condition which would place the individual at elevated risk of serious COVID-19 infection, or any other factor which may make the individual eligible for priority COVID-19 vaccination (i.e. ahead of others in their age group).
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, including IRVs e.g. amphotericin B, chlortetracycline, neomycin, polymyxin, streptomycin
* Any history of anaphylaxis in relation to vaccination.
* Clinically significant laboratory abnormality as judged by the PI or other delegated individual.
* Receipt of any previous rabies vaccinations, including an incomplete course.
* History of vaccination with previous adenoviral vectored vaccines in the 6 months prior to enrolment in the study, or of vaccination with any other vaccine (including non-adenovirus-vectored COVID-19 vaccines) in the 28 days prior to enrolment.
* Planned / likely receipt of any other vaccine within 28 days after enrolment.
* History of bleeding disorder (e.g., factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture, or continuous anticoagulation e.g., with warfarin
* History of confirmed major thrombotic event, (including cerebral venous sinus thrombosis, deep vein thrombosis, pulmonary embolism) or,
* History of antiphospholipid syndrome.
* History of prior receipt of unfractionated heparin
* History of heparin induced thrombocytopenia
* Receipt of any blood products/ immunoglobulins within the three months preceding the planned administration of the vaccine candidate.
* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period.
* Seropositive for hepatitis B surface antigen (HBsAg) or hepatitis C (HCV IgG).
* Likelihood of travel away from the study area.
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Any other significant disease, disorder or situation which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Contraindication to use of paracetamol

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 174 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Safety profile of ChAdOx2 RabG in healthy adult volunteers (18-45 years) and young children (2-6 years) residing in a rabies-endemic country assessed by the occurrence of solicited adverse events. | Assessment of solicited AEs in the first 7 days post vaccination
  Occurrence of solicited local and systemic adverse events (i.e: pain, redness, swelling and pruritus at injection site and temperature, feverishness, myalgia, arthralgia, malaise, headache, fatigue and nausea).
Safety profile of ChAdOx2 RabG in healthy adult volunteers (18-45 years) and young children (2-6 years) residing in a rabies-endemic country assessed by the occurrence of solicited adverse events. | Unsolicited AEs to be assessed up to 28 days post vaccination
  Occurrence of unsolicited local and systemic adverse events
Safety profile of ChAdOx2 RabG in healthy adult volunteers (18-45 years) and young children (2-6 years) residing in a rabies-endemic country assessed by the occurrence of solicited adverse events. | SAEs will be collected from enrolment until the end of the follow-up period (Day 1839)
  Occurrence of serious adverse events
Safety profile of ChAdOx2 RabG in healthy adult volunteers (18-45 years) and young children (2-6 years) residing in a rabies-endemic country assessed by the occurrence of solicited adverse events. | Clinical Laboratory AEs to be assessed up to 28 days post vaccination
  Occurrence of laboratory adverse events defined as clinically significant changes from baseline. Haematology (Full Blood Count) and Biochemistry (Kidney and Liver Function Tests) will be assessed.

SECONDARY OUTCOMES:
Immunogenicity of ChAdOx2 RabG administered to adults and young children residing in a rabies endemic country following primary vaccination, including the length of response maintenance, and secondary (recall) response. | At Days 0, 28, 56, 186, 365, 730, 1095, 1460, 1825
  Rapid fluorescent focus inhibition test (RFFIT) of rabies virus neutralising antibody
Comparison of immunogenicity of ChAdOx2 RabG with a single visit two site intradermal IRV PrEP regimen | At days SPEP+0 and SPEP+7
  Anamnestic rabies virus neutralising antibody response as assessed by rapid fluorescent focus inhibition test (RFFIT), at 7 days following simulated rabies virus exposure through IRV administration

CONTACTS AND LOCATIONS:
Overall Officials: Alexander D Douglas, Principal Investigator — Jenner Institute
Locations (1):
- IHI Clinical Trial Facility, Bagamoyo, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be made available on direct request to the Principal Investigator. Proposals will be reviewed by the sponsor, Principal Investigator, and collaborators on the basis of scientific merit. Data will be shared following approval of the proposal and signed data-access agreements.
Supporting Information: Study Protocol, SAP, ICF